CLINICAL TRIAL: NCT05390801
Title: Congenital Aniridia Patient Questionnaire
Acronym: Aniridia-Quizz
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220119; 2021-A02363-38 (Other: ID-RCB Number)
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Congenital Aniridia
Keywords: Congenital aniridia; Patient survey; Patients knowledge
MeSH Terms: conditions — Aniridia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Any patient ≥ 18 years old with congenital aniridia, able to respond independently to a questionnaire and patients under 18 years old with congenital aniridia, whose parents can respond for their child.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey developed by ophthalmologists from the Ophthalmology Department of the Necker-Enfants Malades Hospital, fill out only once by patients with congenital aniridia in order to identify eye and systemic manifestations in congenital aniridia and to determine the patients' knowledge of their own disease.

SUMMARY:
Congenital aniridia is a pan-ocular genetic disease characterized by a partial or complete absence of the iris, hence its name. The prevalence ranges from 1 / 40,000 to 1 / 96,000 births, but it may be underestimated. This condition combines several types of eye damage and could associate systemic manifestations, with a variable phenotype and genotype.

This study aims to identify eye and systemic manifestations in congenital aniridia and to determine the patients' knowledge of their own disease through a survey prepared by ophthalmologists from the Ophthalmology Department of Necker-Enfants Malades Hospital, reference center in France for this pathology. The patient fills it out only once.

DETAILED DESCRIPTION:
Congenital aniridia is a pan-ocular genetic characterized by partial or complete absence of the iris, hence its name. The prevalence ranges from 1 / 40,000 to 1 / 96,000 births, but it may be underestimated. This condition combines several types of eye damage :

* Partial or complete absence of iris, iris abnormalities
* Glaucoma
* Cataract
* Corneal opacifications with neovascularization
* Foveal hypoplasia with nystagmus
* Hypoplasia of the optic nerve The signs of the disease vary from one individual to another, even within the same family. Iris abnormalities and foveolar hypoplasia are the most constant signs. Affected patients have a highly compromised visual prognosis in adulthood, and are very often considered visually impaired with criteria for legal blindness.

Congenital aniridia can also be associated with several severe systemic manifestations, including syndromic aniridia (WAGR syndrome and Gillespie syndrome).

The major gene responsible for autosomal dominant forms of congenital aniridia is PAIRED BOX GENE 6 (PAX6) (MIM#607108) with over 500 pathogenic variants reported to date.

Congenital aniridia is therefore a rare, pan-ocular disease associating systemic manifestations, with a variable phenotype and genotype.

This study aims to identify eye and systemic manifestations in congenital aniridia and to determine the patients' knowledge of their own disease through a survey prepared by ophthalmologists from the Ophthalmology Department of Necker-Enfants Malades Hospital, reference center in France for this pathology. The patient fills it out only once.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥ 18 years old with congenital aniridia and able to respond independently to the study survey,
* or patients under 18 years old with congenital aniridia, whose parents can answer the study survey,
* adult patients or holders of parental authority and minor patients informed and not opposed to participation in the study.

Exclusion Criteria:

- Patients with neurological disorders preventing them from answering the survey, except in the case of minor patients, if the parents can answer for the patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed in Necker Enfants Malades hospital, the referral center in France for congenital aniridia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Ocular and systemic manifestations in congenital aniridia | 24 months
  To identify eye and systemic manifestations in congenital aniridia through a survey prepared by ophthalmologists. The answers of the survey will be compared with data from the patient's medical file.

SECONDARY OUTCOMES:
Patient's autonomy | 24 months
  Descriptive analysis of the patient's answers and data from the patient's medical file to determine the impact of the disease on patient's autonomy.
  Questions in the survey concerning patient's autonomy will be compared to the data collected in the medical file. For instance: help with activities of daily living, computer/phone use, lifestyle, outdoor and indoor travel, etc.
Patients knowledge | 24 months
  Descriptive analysis of the patient's answers and data from the patient's medical file to determine how well patients know their disease and potential complications.
  Questions in the survey concerning the etiology, complications and evolution of the disease will be compared with the data collected in the medical file in order to determine the degree of knowledge of the patients of the disease.
Factors influencing patient knowledge | 24 months
  To determine the influence of factors such as age, sex, origin and profession on patients' knowledge of their disease according to survey answers.
Parental knowledge | 24 months
  Descriptive analysis of the parents' answers and data from the patient's medical file to determine parents' knowledge of their child's disease and potential complications.
  For patients < 18 years old, the parents' answers of the questions in the survey concerning the etiology, complications and evolution of the disease will be compared with the data collected in the medical file.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Daruich, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Dominique Bremond-Gignac, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No